CLINICAL TRIAL: NCT05727137
Title: Analgesic Efficacy of Daily Single Shot Adductor Canal Block Versus Continuous Adductor Canal Block After Total Knee Arthroplasty
Brief Title: Daily Single Shot Adductor Canal Block Versus Continuous Adductor Canal Block After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University (Other)
Responsible Party: Principal Investigator, Seokha Yoo, Clinical assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2209-136-1362
Record Dates: First submitted 2023-01-25; First posted 2023-02-14 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single shot adductor canal block (Experimental)
  Interventions: Procedure: Single shot adductor canal block
- Continuous adductor canal block (Active Comparator)
  Interventions: Procedure: Continuous adductor canal block

INTERVENTIONS:
Procedure: Single shot adductor canal block — Single shot adductor canal block on the the first and second postoperative day.
  Arms: Single shot adductor canal block
Procedure: Continuous adductor canal block — A catheter will be placed in the adductor canal and connected to a continuous patient-controlled analgesia pump.
  Arms: Continuous adductor canal block

SUMMARY:
This study will compare the analgesic efficacy of daily single-shot adductor canal block(ABC) versus continuous ACB after total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
Patients 19-75 years old, of ASA classification I-III scheduled for unilateral TKA, will be enrolled and randomized into two groups, single-shot ACB group and continuous ACB group. In both groups, participants will be administered a single-shot ACB immediately after the end of the operation. The single-shot ACB group will receive two separate single-shot ACBs, on the first and second postoperative day. A nerve block catheter will be placed in patients in the continuous ACB group, which will be connected to a patient-controlled analgesia pump until the second postoperative day. The primary outcome of this study is the average NRS pain score at rest from the end of surgery to 2 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I, II, III
* Patients scheduled for unilateral knee arthroplasty

Exclusion Criteria:

* Anesthesia other than spinal anesthesia
* Chronic opioid use
* Uncontrolled diabetes of HbA1c>7.5
* Neuromuscular pathology of the ipsilateral leg
* Second-look knee arthroplasty
* Inability to communicate (e.g. dementia)
* Hypersensitivity to ropivacaine
* BMI > 40
* Pregnancy

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Average NRS pain score at rest | first 48h after end of surgery
  average of numerical rating scale (0: no pain, 10: worst imaginable pain) pain scores from 8 time points during 48h (+4h, +8h, +12h from end of surgery, 6AM, 2PM, 10PM of postoperative day 1, and 6AM and 2PM of postoperative day 2)

SECONDARY OUTCOMES:
numerical rating scale (0: no pain, 10: worst imaginable pain) pain score at rest at +4h from end of surgery | +4h from end of surgery
numerical rating scale (0: no pain, 10: worst imaginable pain) pain score during movement at +4h from end of surgery | +4h from end of surgery
NRS pain score at rest at +8h from end of surgery | +8h from end of surgery
numerical rating scale (0: no pain, 10: worst imaginable pain) pain score during movement at +8h from end of surgery | +8h from end of surgery
numerical rating scale (0: no pain, 10: worst imaginable pain) pain score at rest at +12h from end of surgery | +12h from end of surgery
numerical rating scale (0: no pain, 10: worst imaginable pain) pain score during movement at +12h from end of surgery | +12h from end of surgery
numerical rating scale (0: no pain, 10: worst imaginable pain) pain score at rest at 6AM on postoperative day 1 | 6AM on postoperative day 1
numerical rating scale (0: no pain, 10: worst imaginable pain) pain score during movement at 6AM on postoperative day 1 | 6AM on postoperative day 1
NRS pain score at rest at 2PM on postoperative day 1 | 2PM on postoperative day 1
NRS pain score during movement at 2PM on postoperative day 1 | 2PM on postoperative day 1
NRS pain score at rest at 10PM on postoperative day 1 | 10PM on postoperative day 1
numerical rating scale (0: no pain, 10: worst imaginable pain) pain score during movement at 10PM on postoperative day 1 | 10PM on postoperative day 1
numerical rating scale (0: no pain, 10: worst imaginable pain) pain score at rest at 6AM on postoperative day 2 | 6AM on postoperative day 2
NRS pain score during movement at 6AM on postoperative day 2 | 6AM on postoperative day 2
numerical rating scale (0: no pain, 10: worst imaginable pain) pain score at rest at 2PM on postoperative day 2 | 2PM on postoperative day 2
numerical rating scale (0: no pain, 10: worst imaginable pain) pain score during movement at 2PM on postoperative day 2 | 2PM on postoperative day 2
Posteoperative opioid administration in morphine equivalents | from end of surgery to 48h after surgery
Incidence of catheter tip dislocation | at 2PM on postoperative day 1 and 2
  The catheter tip is considered to be dislocated if the catheter tip is located outside the adductor canal
Incidence of extravasation from catheter insertion site | at 2PM on postoperative day 1 and 2
Incidence of sleep disturbance due to pain | from end of surgery to postoperative day 2
Incidence of numbness of anterior thigh area | at 2PM on postoperative day 1 and 2
Strengh of quadratus femoris muscle (unit: kgf) | at 2PM on postoperative day 1 and 2
Incidence of falls during hospital stay | from end of surgery to 48h after surgery
Postoperative range of motion of knee joint | at 2PM on postoperative day 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Seokha Yoo, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim H, Yoo S, Kwon S, Kim Y, Bae J, Kim YJ, Cho YJ, Kim JT, Lim YJ. Analgesic Efficacy of Repeated Daily Injections Versus Continuous Adductor Canal Block After Total Knee Arthroplasty: An Open-Label, Randomized Clinical Trial. Anesth Analg. 2026 Jan 1;142(1):132-139. doi: 10.1213/ANE.0000000000007427. Epub 2025 Feb 18. PMID 39964911